CLINICAL TRIAL: NCT06329154
Title: Clinical Study On Extracorporeal Shock Wave Therapy For Rotator Cuff Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Liu, MD (Other)
Responsible Party: Sponsor-Investigator, Yong Liu, MD, chief physcician, The First Affiliated Hospital of Dalian Medical University
Organization: The First Affiliated Hospital of Dalian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PJ-KS-KY-2024-03(X)
Record Dates: First submitted 2024-03-06; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Rotator Cuff Injuries
Keywords: Rotator Cuff Injuries; Extracorporeal Shockwave Therapy
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: assessor was blinded. The assessor, who not participated in the study, was experienced, and well qualified in the use.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extracorporeal shock wave therapy group (Experimental): The experimental group received extracorporeal shock wave therapy combined with conventional rehabilitation therapy. Conventional rehabilitation therapy includes medium frequency electricity, ultrasound, ultrashort wave, laser, wax therapy, etc.
  Interventions: Device: Extracorporeal shock wave therapy
- control group (Active Comparator): The control group received conventional rehabilitation therapy. Conventional rehabilitation therapy includes medium frequency electricity, ultrasound, ultrashort wave, laser, wax therapy, etc.
  Interventions: Other: conventional rehabilitation therapy

INTERVENTIONS:
Device: Extracorporeal shock wave therapy — The experimental group received extracorporeal shock wave therapy combined with conventional rehabilitation therapy. The control group was only given conventional rehabilitation therapy. According to the patient's tolerance and the specific condition, extracorporeal shock wave therapy was performed twice a week, 2000-3000 times each time, energy parameters of 2.5-3.5Bar, 8-15Hz, treatment interval > 1 day, consecutive 4 weeks. Conventional rehabilitation therapy included medium frequency electricity, ultrasound, ultrashort wave, laser and wax therapy. Routine rehabilitation was given once a day, 5 times a week for 4 weeks.
  Arms: extracorporeal shock wave therapy group
Other: conventional rehabilitation therapy — Conventional rehabilitation therapy included medium frequency electricity, ultrasound, ultrashort wave, laser, and wax therapy (same as the control group). Routine rehabilitation was given once a day, 5 times a week for 4 weeks.
  Arms: control group

SUMMARY:
This clinical trial aims to learn about the effect of extracorporeal shock wave therapy on rotator cuff injuries. The main question it aims to answer is the efficacy of extracorporeal shock wave therapy on the improvement of pain, shoulder function, and quality of life in patients with rotator cuff injuries. The experimental group of patients received extracorporeal shock wave therapy combined with conventional rehabilitation therapy. The control group only received conventional rehabilitation therapy. Compare the two groups to explore the therapeutic effect of extracorporeal shock wave therapy on rotator cuff injuries.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of rotator cuff injuries in 2019 American Academy of Orthopaedic Surgeons Clinical Practice Guideline for rotator Cuff Injuries (diagnostic criteria: （1）The clinical signs included positive empty cup test and full cup test, positive internal rotation resistance test in abduction and external rotation position and positive Jobe sign in lateral position. (2) Imaging: magnetic resonance imaging, magnetic resonance arthrography or ultrasound showed rotator cuff injuries, including supraspinatus, infraspinatus, teres minor and subscapularis tendon injuries);
* Definite imaging diagnosis: magnetic resonance imaging, magnetic resonance arthrography or ultrasound examination;
* The shoulder joint did not receive surgical treatment;
* Both sexes, aged 20-80 years old;
* Stable vital signs, good communication, and active cooperation to complete the relevant evaluation and treatment;
* Informed consent was obtained from patients or their families before treatment.

Exclusion Criteria:

* MRI showed medium, large and huge full-thickness rotator cuff tears;
* Skin damage or skin disease at the application site;
* Previous history of shoulder surgery;
* Pregnant or lactating women;
* Allergic constitution;
* Patients with primary diseases of the heart, liver, kidney, or hematopoietic system, patients with mental disorders, patients with built-in cardiac pacemaker, and patients with implanted metal medical devices;
* complicated with other diseases that cause body pain;
* Unable to cooperate with the completion of the whole treatment and follow-up.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-01-27 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Visual Analogue Scale at 4 weeks | baseline and 4 weeks
  Visual analogue Scale is the most commonly used single-dimensional measurement of pain intensity. The scale mainly consists of a 10-cm straight line, one end of which indicates "no pain at all" and the other end indicates "the most severe pain imaginable" or "pain to the extreme" etc. The patient will be asked to mark the corresponding position on this line to represent the intensity of the pain they feel at that time.
Change from Baseline Range of Motion at 4 weeks | baseline and 4 weeks
  The range of motion of the shoulder joint refers to the active and passive range of motion of the shoulder joint measured with a protractor, including forward flexion, back extension, abduction, internal rotation, and external rotation.
Change from Baseline Constant-Murley Score at 4 weeks | baseline and 4 weeks
  Constant-Murley Score is the unified shoulder score of the European Society for Shoulder and Elbow Surgery. The left and right shoulder joints were scored separately. It mainly includes 8 aspects of shoulder joint-related problems: 1, pain; 2. Degree of influence on daily life; 3. The hand can lift the height that can be reached; 4. Upper limb abduction muscle strength; 5. The degree of upper limb forward lifting; 6, the degree of upper limb abduction; 7. The degree of external rotation of the upper limbs; 8, the degree of internal rotation of the upper limb can be achieved.
Change from Baseline Isokinetic muscle strength testing at 4 weeks | baseline and 4 weeks
  Isokinetic muscle testing can be used for quantitative measurement of muscle strength, and the evaluation results have objectivity, accuracy, repeatability, and high sensitivity.
Change from Baseline Magnetic resonance imaging at 4 weeks | baseline and 4 weeks
  Magnetic resonance imaging has good soft tissue resolution and can clearly show the injuries of tendons and ligaments around the shoulder joint. It is one of the main examination methods for the evaluation of rotator cuff injuries.
Change from Baseline Musculoskeletal ultrasound at 4 weeks | baseline and 4 weeks
  Musculoskeletal ultrasound uses high-frequency ultrasound to diagnose musculoskeletal diseases, which can clearly show the superficial soft tissue structures such as muscles, tendons, ligaments, peripheral nerves, and their lesions. It is one of the main examination methods for the evaluation of rotator cuff injuries.

SECONDARY OUTCOMES:
Change from Baseline American Shoulder and Elbow Surgeons Score at 4 weeks | baseline and 4 weeks
  Developed by the American Society of Shoulder and Elbow Surgeons, it measures shoulder pain, function, or disability. The pain and function subscales each account for 50 points, and the total score ranges from 0 to 100, with higher scores indicating better conditions, i.e. less severe symptoms; The lower the score, the more severe the disease. The assessment consisted of 1 item for pain and 10 items for function.
Change from Baseline Shoulder Pain and Disability Index at 4 weeks | baseline and 4 weeks
  The Shoulder Pain and Disability Index measures the pain and disability associated with shoulder lesions. It consists of two subscales: pain and functional or disability. The total score is converted to a score of 0 to 100, with higher scores indicating greater pain and disability.
Change from Baseline Disability of the Arm, Shoulder and Hand Score at 4 weeks | baseline and 4 weeks
  The Disability of the Arm, Shoulder, and Hand Score was developed by the American Academy of Orthopaedic Surgeons and the Institute for Work and Health to measure the level of upper extremity-related symptoms, function, or disability. There were 30 items: 5 symptom related and 25 function related. The total score is converted to a 0-100 percentage, with higher scores indicating greater disability. Another two subscales can be selected: work and exercise.
Change from Baseline University of California at Los Angeles Shoulder Scale at 4 weeks | baseline and 4 weeks
  The University of California at Los Angeles Shoulder Scale was developed by Dr. Amstutz and colleagues at the University of California at Los Angeles Shoulder Scale. Pain, function, active forward flexion, strength of forward flexion, and total satisfaction. The total score ranges from 0 to 35, and some studies will convert the score into a score of 0 to 100, with higher scores indicating better conditions.
Change from Baseline Pittsburgh sleep quality index at 4 weeks | baseline and 4 weeks
  The Pittsburgh sleep quality index was developed by Dr. Buysse, a psychiatrist at the University of Pittsburgh in 1989. It was used to assess the sleep quality of the subjects in the last month. It consisted of 19 self-rated items and 5 other-rated items, of which the 19th self-rated item and 5 other-rated items were not involved in the scoring. The total score of each component was the total score. The total score ranged from 0 to 21, and the higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China